CLINICAL TRIAL: NCT01882218
Title: A Comparison of Direct Peritoneal Resuscitation Plus Conventional Resuscitation Versus Conventional Resuscitation Alone in Patients Undergoing Hepatic Resection for Cancer
Brief Title: Direct Peritoneal Resuscitation Plus Conventional Resuscitation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not feasable at this site
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Jason Smith, MD, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12.0262
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Hepatic Cancer
Keywords: Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Galactose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Standard liver surgery and post-operative treatment
  Interventions: Drug: Standard Treatment
- Galactose (Experimental): Standard liver surgery with direct peritoneal resuscitation with galactose after surgery.
  Interventions: Drug: Galactose

INTERVENTIONS:
Drug: Galactose — After surgery, galactose will be dripped into the belly for up to 24 hours after surgery
  Arms: Galactose
Drug: Standard Treatment — Standard liver surgery.
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to find out if direct peritoneal resuscitation (DPR) (putting a sugar solution into the abdominal cavity) helps blood flow through vital organs in the body that may suffer from low blood flow due to surgery. We will also try to find out if the DPR will help patients recover faster from liver surgery. Lastly, this study will also try to find if direct peritoneal resuscitation decreases levels of signaling chemicals in the blood called 'cytokines' and a protein called high-mobility group protein 1, which is known to cause tissue damage.

DETAILED DESCRIPTION:
Our study will focus on 108 patients requiring hepatic resection for colorectal cancer metastasis or primary hepatocellular carcinoma. These patients will then be randomized into two 54 patient arms: the control arm of conventional resuscitation only and the experimental arm of conventional resuscitation with DPR immediately post operatively. Patient exclusion criteria will be: 1) unable to obtain proper consent for enrollment, 2) age less than 18 years or greater than 75 years, 3) chronic renal failure, cirrhosis, or congestive heart failure, 4) patients requiring portal venous embolization prior to resection, or 5) women who are pregnant or lactating/breast feeding. A pregnancy test (urine or blood) will be done for female subjects of child bearing potential the day prior or the morning of surgery per the usual standard of care pre-op labs.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer
* Scheduled for liver resection
* 18 to 75

Exclusion Criteria:

* Chronic renal failure
* Cirrhosis
* Congestive heart failure
* Requiring portal venous embolization prior to resection
* Pregnant or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Morbidity | Six months

SECONDARY OUTCOMES:
Cytokine levels | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Smith, MD, Principal Investigator — U Louisville
Locations (2):
- United States (2):
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No